CLINICAL TRIAL: NCT03780881
Title: Worse Than Expected - Differences Between Healthy and Depressed People in Processing Unexpectedly Negative Information
Brief Title: EXperimental Paradigm to Investigate Expectation Change in Depression 4
Acronym: EXPECD4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2018-37k
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two experimental groups in parallel for the duration of the study
Who Masked: Investigator
Masking Description: The investigator randomly assigns participants to one of the experimental conditions. Participants are not aware which experimental condition they are allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expectation confirmation (Experimental): The participants in this group receive manipulated feedback indicating that their performance was very good in the test they had previously worked on. This feedback is intended to confirm the previously induced positive expectations of their own performance.
  Interventions: Behavioral: Expectation confirmation
- Expectation disconfirmation (Experimental): The participants in this group receive manipulated feedback indicating that their performance was below average in the test they had previously worked on. This feedback is intended to negatively disconfirm the previously induced positive expectations of their own performance.
  Interventions: Behavioral: Expectation disconfirmation

INTERVENTIONS:
Behavioral: Expectation confirmation — Participants receive manipulated feedback indicating that their performance was above average in the test they had previously worked on. This feedback is intended to confirm the previously induced positive expectations of their own performance.
  Arms: Expectation confirmation
Behavioral: Expectation disconfirmation — Participants receive manipulated feedback indicating that their performance was below average in the test they had previously worked on. This feedback is intended to negatively disconfirm the previously induced positive expectations of their own performance.
  Arms: Expectation disconfirmation

SUMMARY:
Research has shown that people with depressive symptoms maintain negative expectations even if they have positive experiences that contradict their expectations. Healthy people, however, change their expectations after unexpected positive experiences. In this experimental study, it will now be examined whether there are also differences between healthy people and people with depressive symptoms in dealing with unexpected negative experiences.

DETAILED DESCRIPTION:
Research has already shown that people with depressive symptoms continue to hold on to negative expectations even if they have positive experiences that contradict their expectations. By contrast, healthy people change their expectations after unexpectedly positive experiences. In this experimental study, the authors will now examine whether there are also differences between healthy people and people with depressive symptoms in processing unexpectedly negative experiences. It is hypothesized that people with depressive symptoms change their expectations in a negative direction after unexpectedly negative experiences, while healthy people continue to hold on to an optimistic view.

ELIGIBILITY:
Inclusion Criteria (clinical sample):

* diagnosis of major depression
* at least 18 years old
* sufficient German language skills

Exclusion Criteria (clinical sample):

* participation in previous studies on changes in expectations

Inclusion Criteria (healthy sample):

* at least 18 years old
* sufficient German language skills

Exclusion Criteria (clinical sample):

* participation in previous studies on changes in expectations
* current diagnosis of any mental disorder
* diagnosis of major depression in the past
* currently receiving psychotherapeutic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2018-11-11 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
2-Item Performance Expectations Scale - generalized | Immediately before the performance test and immediately after completion of the performance test
  Changes from baseline to postassessment in generalized performance expectations. Each item is scored from 1 to 7 (1 = very negative expectations, 7 = very positive expectations), yielding a total score between 2 and 14. Higher total scores reflect more positive expectations.

SECONDARY OUTCOMES:
2-Item Performance Expectations Scale - task-specific | Immediately before the performance test and immediately after completion of the performance test
  Changes from baseline to postassessment in task-specific performance expectations. Each item is scored from 1 to 7 (1 = very negative expectations, 7 = very positive expectations), yielding a total score between 2 and 14. Higher total scores reflect more positive expectations.

OTHER OUTCOMES:
5-Item Cognitive Immunization after Performance Feedback (CIPF) scale | Immediately after completion of the performance test
  Engagement in cognitive immunization strategies after receiving performance feedback. Each item is scored from 1 to 7 (1 = no cognitive immunization, 7 = great engagement in cognitive immunization), yielding a total score between 5 and 35. Higher total scores reflect a greater engagement in cognitive immunization strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kube, PhD, Principal Investigator — Philipps University Marburg
Locations (1):
- Schoen Klinik Bad Arolsen, Bad Arolsen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared